CLINICAL TRIAL: NCT02474849
Title: A Pharmacokinetic Study to Compare Nicotine Delivery From e Cigarettes and a Conventional Cigarette in Healthy Subjects During a Brief Period of ad Libitum Use
Brief Title: Pharmacokinetic Study Comparing Nicotine Delivery From E-cigarettes and a Conventional Cigarette in Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: British American Tobacco (Investments) Limited (Industry)
Collaborators: LA Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BAT4215006
Record Dates: First submitted 2015-06-11; First posted 2015-06-18 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Conventional cigarette (Active Comparator)
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette
- First-generation e-cigarette (Experimental)
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette
- Rechargeable cig-like e-cigarette (Experimental)
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette
- Closed modular system e-cigarette A (Experimental)
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette
- Closed modular system e-cigarette B (Experimental)
  Interventions: Other: Use electronic cigarette or smoke conventional cigarette

INTERVENTIONS:
Other: Use electronic cigarette or smoke conventional cigarette — Use of electronic cigarette or smoking conventional cigarette ad libitum for 5 minute period

SUMMARY:
This study will compare nicotine delivery, heart rate, puffing parameters and product satisfaction in healthy subjects either using several different types of electronic cigarettes or smoking a conventional cigarette.

ELIGIBILITY:
Inclusion Criteria:

1. Prior to study start, subjects must be daily users of newer generation e-cigarette devices which they have used regularly for a minimum of three months. The solutions used in their e-cigarettes must contain nicotine. Subjects must also be occasional smokers of combustible cigarettes (lower limit of 1 cigarette per month; upper limit of 5 cigarettes per week). Product use status will be confirmed with a urinary cotinine level of ≥200ng/ml (determined using NicAlert cotinine test kit) at screening.
2. Subjects will be males or non-pregnant, non-lactating females, and between 21 and 55 years of age inclusive. Age verification will be performed by checking of Federal or state-issued ID (e.g. passport or driving licence) during screening.
3. Women of child-bearing potential should be using one of the following acceptable methods of contraception : combined (oestrogen and progestogen containing) oral, intravaginal or transdermal hormonal contraception associated with inhibition of ovulation; progestogen-only hormonal contraception, either oral, injected or implanted, associated with inhibition of ovulation; progestogen-only oral hormonal contraception where inhibition of ovulation is not the primary mode of action; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; male or female condom with or without spermicide; cap, diaphragm or sponge with spermicide.
4. Women of non-childbearing potential may be included if they are either surgically sterile (hysterectomy and/or oophorectomy) or postmenopausal for more than 1 year and must have a negative urine pregnancy test result during screening. Women who are surgically sterile must provide documentation of the procedure by an operative report.
5. Male subjects must use an approved method of birth control during the entire study. These subjects must not donate sperm during this time.
6. Subjects must be in good health as determined by medical history, vital signs, blood biochemistry, haematology, urinalysis and physical examination.
7. Subjects must have a body mass index (BMI) between 18 and 30 kg/m2 inclusive. Male subjects must have a weight between 60 and 120kg and female subjects between 50 and 100kg.
8. No clinically significant abnormalities in blood pressure values.
9. Subjects will have negative results for the urinary drug of abuse screening and ethanol test.
10. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.

To be confirmed during each clinic visit:

1. Abstinence from tobacco and nicotine products will be confirmed by an exhaled breath CO reading <10ppm.

Exclusion Criteria:

1. Subjects who have a history of, or clinically active significant, neurological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological disease or other major disorders.
2. Subjects with significant allergies who in the opinion of the Principal Investigator should not be included.
3. Subjects who have been diagnosed with urticaria (hives) or asthma.
4. Persons who have a history of urticaria (hives) in response to any product.
5. Subjects with a recent history of or current drug or alcohol abuse who in the opinion of the Investigator should not be included. Excessive intake of alcohol within the last 6 months, defined as a regular maximum weekly intake of greater than 7 drinks for women or 14 drinks for men. One drink is defined as one pint of regular beer (5% alcohol), 200 ml of wine (12% alcohol), or 25 ml of distilled spirits (40% alcohol).
6. Subjects with an inability to communicate well with the Investigator/study staff (i.e., language problem, poor mental development or impaired cerebral function).
7. Subjects who are participating in another clinical research study or who have participated in a clinical research study in the last 3 months.
8. Subjects who have had treatment with prescription medications within 21 days or over-the-counter medication within 24 hours of the planned first product use occasion, except for those stated in the Inclusion Criteria. For all subjects, prescribed use of blood pressure (beta blockers) and lipid lowering (statin) medications are permitted.
9. Subjects who have used any drugs or substances (except tobacco) known to be strong inducers or inhibitors of any CYP enzymes (formerly known as cytochrome P450 enzymes) within a 28 days period prior to first product administration. For a list of such drugs and substances, please refer to http://medicine.iupui.edu/clinpharm/ddis/main-table/.
10. Subjects who have had any treatment with smoking cessation medications (e.g. Bupropion, Chantix or any NRT) within 30 days of the planned first product use occasion.
11. Subjects with any other clinically significant medical history, in the Investigator's opinion, including conditions which might affect drug absorption, metabolism or excretion.
12. Female subjects, who are pregnant or become pregnant during the course of the study.
13. Subjects who have lost or donated more than 450ml of blood within the 3 months preceding the first product administration.
14. Subjects who are currently trying to stop smoking or to stop using e-cigarettes, or considering stopping in the next two months.
15. Subjects who are unwilling or unable to comply with the study requirements.
16. Subjects who in the opinion of the Investigator should not participate in the study for any other reason.

To be re-confirmed during each clinic visit:

1. Subject continues to meet all screening exclusion criteria.
2. Receipt of any medication since screening visit that may have an impact on the safety and objectives of the study (at the Principal Investigator's discretion).

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Plasma nicotine concentration (Cmax) | -5, 1, 3, 5, 6, 7, 9, 15, 40, and 60 minutes relative to the first puff on the cigarette/e-cigarette
  Nicotine pharmacokinetics
Plasma nicotine concentration (Tmax) | -5, 1, 3, 5, 6, 7, 9, 15, 40, and 60 minutes relative to the first puff on the cigarette/e-cigarette
  Nicotine pharmacokinetics
Plasma nicotine concentration (AUC0-60) | -5, 1, 3, 5, 6, 7, 9, 15, 40, and 60 minutes relative to the first puff on the cigarette/e-cigarette
  Nicotine pharmacokinetics

SECONDARY OUTCOMES:
Change in heart rate | 5 minutes before, during, and 5 minutes after puffing period
  Pharmacodynamics
Number of puffs taken | During 5 minute ad libitum puffing period
Duration of puffs taken | During 5 minute ad libitum puffing period
Subjective measurement of product satisfaction | After 5 minute product use period

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Nides, PhD, Principal Investigator — Los Angeles Clinical Trials
Locations (1):
- Los Angeles Clinical Trials, Burbank, California, United States